CLINICAL TRIAL: NCT06125314
Title: A Multicenter, Non-Interventional, Retrospective Study Aims to Estimate the Prevalence and Describe the Clinical Manifestations of HER2-Low Breast Cancer Reported in Unresectable and/or Metastatic Breast Cancer Patients Who Progress on Anti-Cancer Therapy Identified as HER2- Negative From Patient Medical Records in The Gulf Council Cooperation Region
Brief Title: HER2 TREAT Study: Retrospective Study to Estimate the Prevalence of HER2-low in Unresectable and/or Metastatic Breast Cancer Patients Who Progress on Anti-Cancer Therapy Identified as HER2-Negative From Patient Medical Records in The Gulf Cooperation Council
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00197
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasms; Breast Cancer; Breast Carcinoma; Genes; HER2
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
HER2-low Breast cancer (BC) has emerged as a new subtype of BC with distinct clinical, pathological, and prognostic features. Little is known about the prevalence of the HER2-low subtype in HER2-negative patients, and previous reports showed variations in the criteria used to define the HER2-low subtype. Besides, data on the clinical features and prognosis of HER2-low patients are limited, and it is still unclear whether HER2-low BC has a prognostic value. Identifying the prevalence and clinical features of HER2-low BC can help establish a more accurate and reproducible definition of HER2-low BC. In the Gulf Cooperation Council (GCC) region, BC is the most common malignancy in women and still poses a significant burden on healthcare resource utilization, moreover, there is only one record for reimbursed HER2 IHC status, categorized as HER2-positive and HER2-negative. It is important to understand the prevalence, clinical features, and outcomes of HER2-low in BC patients from the GCC In this retrospective, non-interventional, multicenter study, the aim to describe the prevalence of HER2-low BC among the current HER2-negative BC population using rescored HER2 IHC samples. The local treatment patterns and the outcomes will be analyzed using the information abstracted from the corresponding medical chart review. The study will cover the GCC region countries (United Arab Emirates [UAE], Saudi Arabia, Qatar, Kuwait, and Oman)

ELIGIBILITY:
Inclusion Criteria:

* women ≥ 18 years of age at date of diagnosis
* Patients must have a histological or cytological confirmed diagnosis of Unresectable or/and mBC between 01st January 2018 and 31st December 2022.
* Patients with at least 12 months of follow-up data (from the index date) in the medical records at the participating site unless patient died.
* Patients must have been diagnosed as HER2-negative (HER2 IHC 0, 1+, 2+/ISH-), regardless of hormone status.
* Patients who are diagnosed and/or progressed on at least one prior systemic anticancer therapy (e.g., ET, chemotherapy, CDK4/6i, targeted therapies other than anti- HER2, or immunotherapy) in the metastatic setting.
* Patients must have historical HER2 fixed tissue IHC stained slides in acceptable quality to allow retesting of HER2 expression only in case of the absence of accurate scoring of IHC/ISH in pathology report.

Exclusion Criteria:

* Have a history of other malignancies other than basal cell carcinoma of the skin and squamous cell carcinoma of the skin.
* Patients who are HER2 positive (with historical HER2 status of IHC 2+/ISH+ or 3+, or HER2 amplified.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult (aged > 18 years old) patients with a confirmed diagnosis of HER2-negative (assessed preferably by Ventana 4b5 assay) Unresectable and/or mBC who presented to the participating centers within the period from 1st January 2018 to 31st December 2022 and who are diagnosed and/or progressed on at least one prior systemic anti-cancer therapy (Endocrine therapy, chemotherapy, CDK4/6i, targeted therapies other than anti-HER2, or PDL1 inhibitor) , regardless of their hormonal status.
Sampling Method: Non-Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
HER2-low prevalence based on rescoring of historical HER2 fixed tissue slides among HER2-negative Unresectable or/and metastatic Breast Cancer patients. | 1st January 2018 to 31st December 2022

CONTACTS AND LOCATIONS:
Locations (7):
- Research Site, Kuwait City, Kuwait
- Research Site, Doha, Qatar
- Saudi Arabia (2):
  - Research Site, Mecca, Saudi Arabia
  - Research Site, Riyadh
- United Arab Emirates (3):
  - Research Site, Abu Dhabi
  - Research Site, Al Ain City
  - Research Site, Dubai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133FR00197&attachmentIdentifier=1362f3de-28aa-40df-8b26-9b217a97a9ea&fileName=CSR_synopsis_redacted.pdf&versionIdentifier=